CLINICAL TRIAL: NCT02661139
Title: Prospective Registry of Prosthodontic Rehabilitation in Oncology Patients Undergoing Jaw Reconstruction
Acronym: O-BRIDGE
Status: Recruiting | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, Maxillofacial surgeon, Head of Department, AZ Sint-Jan AV
Other Study IDs: B049201525496
Record Dates: First submitted 2016-01-11; First posted 2016-01-22 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Cancer; Osteonecrosis; Osteoradionecrosis
Keywords: bisphosphonates; jaw reconstruction; prosthetic rehabilitation; quality of life; monoclonal antibodies' targeted therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Osteonecrosis; Osteoradionecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to develop a prospective database in which patient demographics, surgical, dental, prosthetic and QOL parameters collected during consecutive visits within the framework of routine practice, are being registered for each oncological patient eligible for (immediate/delayed) fixed prosthodontic rehabilitation at time of oral cavity reconstruction

DETAILED DESCRIPTION:
The number of patients requiring major ablative surgery in the oral cavity, including partial/radical mandibular or maxillary resection, due to a head and neck carcinoma, osteoradionecrosis (ORN), or medication-related osteonecrosis of the jaw (MRONJ) has not been accurately reported. Surgical reconstruction to restore oral function and aesthetics forms a challenge to maxillofacial surgeons, and greatly impacts patient' quality of life (QOL). Recently, an active collaboration between the surgeons of the Oral and Maxillofacial Surgery Unit and the prosthodontist (LB) of the Department of Dentistry at the General Hospital Saint-John Bruges led to the development of the "Oncology-bridge (O-bridge)" protocol, which offers (immediate/delayed) fixed prosthetic rehabilitation in a minimum of sessions and a strongly reduced two-week treatment time, consequently accelerating patient' improved QOL at a considerably reduced cost.

The investigators aim to develop a prospective database in which patient demographics, surgical, dental, prosthetic and QOL parameters collected during consecutive visits within the framework of routine practice, are being registered for each oncological patient eligible for (immediate/delayed) fixed prosthodontic rehabilitation at time of oral cavity reconstruction This could provide the investigators with more information about potential patient, surgical and prosthetic factors influencing short- and long-term biological and mechanical stability, as well as patient QOL. Moreover, registration of those results could function as a measurement of quality of care, and could be used for sample size calculation for future large prospective trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages
* Patients of all genders
* Patients with a histologically or clinically confirmed diagnosis of ORN, MRONJ, as classified by Ruggiero et al. (Ruggiero, et al., 2014) or carcinoma located in the oral cavity and jawbone, requiring segmental or total jaw resection
* Patients eligible for jaw and oral cavity reconstruction combined with immediate/delayed implant loading for fixed prosthetic rehabilitation
* Patients not eligible for conventional removable prosthetic rehabilitation

Exclusion Criteria:

* Patients with a clinically confirmed diagnosis of osteonecrosis not related to an oncological diagnosis or treatment
* Patients with medical contraindications for jaw reconstruction combined with immediate implant loading for fixed prosthetic rehabilitation
* Patients eligible for conventional removable prosthetic rehabilitation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consenting patients with a histologically confirmed oncology diagnosis that requires major ablative surgery of the oral cavity, including segmental or total jaw resection, due to head and neck cancer, ORN or MRONJ
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2013-06; Primary Completion 2022-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
implant survival rate | within 12 months postoperative
bone resorption, as evaluated with cone-beam computed tomography | within 12 months postoperative
prosthesis survival rate | within 12 months postoperative
implant survival rate | within 60 months postoperative
bone resorption, as evaluated with cone-beam computed tomography | within 60 months postoperative
prosthesis survival rate | within 60 months postoperative

SECONDARY OUTCOMES:
Prevalence of oncological patients requiring jaw reconstruction secondary to tumour resection, ORN or MRONJ | within 12 months postoperative
Potential biologic or mechanical risk factors predictive of undesirable functional or aesthetic outcomes, through regression analysis | within 60 months postoperative
Patient' quality of life after prosthetic rehabilitation | until a maximum of 60 months follow-up

OTHER OUTCOMES:
patient satisfaction, as measured through visual analogue scale | until a maximum of 60 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, MD, Principal Investigator — Department of Oral and Maxillofacial Surgery, General Hospital Saint-John Bruges, Bruges, Belgium
Locations (1):
- General Hospital Saint-John Bruges, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No